CLINICAL TRIAL: NCT04533854
Title: SPECTRA: Investigating Signal Change in Malignant and Non-malignant Pleural Effusions and asCitic Fluid Using fTiR Analysis
Brief Title: Investigating Signal Change in Malignant and Non-malignant Pleural Effusions and asCitic Fluid Using fTiR Analysis
Acronym: SPECTRA
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2020/36
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-09

CONDITIONS: Pleural Effusion; Ascites
MeSH Terms: conditions — Pleural Effusion; Ascites

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pleural fluid and ascitic fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is a common cancer, associated with a high mortality rate. Pleural effusions are common in lung cancer, developing in up to 40% of patients. Ascites is common in patients with abdominal malignancies and can be the presenting feature in up to 50% of patients. There is a need for new techniques to improve our diagnostic ability of cancer. FTIR technology could enable a point-of-care test that would provide an initial diagnosis that may determine a change in treatment at the time of the investigation.

DETAILED DESCRIPTION:
Lung cancer accounts for 13% of all new cancer cases in the UK and is the third most common cancer. However, lung cancer has the highest mortality rate, thought partly related to late diagnosis. Pleural effusions develop in up to 40% of patients with lung cancer, and can be the first presenting sign. Current methods of analysing pleural fluid are based on using Light's criteria to distinguish between exudates and transudates depending on the protein and LDH component of the fluid. However, this system does not discriminate between causes of exudative effusions for example malignant effusions vs infective causes. Pleural fluid cytology can identify malignant effusions but gives an average yield of 60% through a labour intensive and time consuming process. If pleural fluid cytology is non-diagnostic, patients require further invasive investigations such as local anaesthetic thoracoscopy, lymph node biopsies or image-guided biopsies to gain a tissue diagnosis. Therefore, determining an alternative, accurate method of diagnosing cancer at the earliest opportunity would reduce the need for further invasive investigations and would provide patients with increased treatment options, thereby increasing survival rates. There are differences in the biochemical composition of malignant and non-malignant effusions thereby offering an opportunity to develop alternative techniques of investigating the cause of these effusions.

Ascites is a common symptom of patients with various underlying cancers; most commonly breast cancer, colon cancer, gastrointestinal cancer and ovarian cancer, and is often associated with significant morbidity. However, up to 50% of patients with malignant ascites present with ascites as the first feature. This symptom is not specific to any type of cancer; current investigations including using serum tumour markers have a low diagnostic specificity and there is a need for new techniques to improve our diagnostic ability.

Fourier transform mid-infrared spectroscopy (FTIR) is a reproducible and relatively simple investigation used to analyse the structural components of tissue or cells. As infrared light is passed through a sample, some light is absorbed and some transmitted through. The resulting signal at the detector presents as a spectrum, representing a 'molecular fingerprint' of the sample. Each chemical structure produces a unique spectral fingerprint making FTIR a useful tool for identifying components of tissue or cells.

Attenuated Total Reflection Linear Variable Filter (ATR-LVF) spectroscopy is a variant of IR spectroscopy in which samples can be examined directly with no preparation needed. ATR-LVF spectroscopy can be performed on benchtop spectrometers with minimal operator training and an immediate result can be obtained.

Both FTIR and ATR-LVF are non-invasive, reproducible, do not damage the sample and have the benefit of only requiring a small sample size to generate results all of which are desirable qualities in developing a new investigation.

FTIR has been used to successfully discriminate between malignant and non-malignant lung tissue6, and also to identify spectral differences in samples of pleural fluid from malignant and non-malignant participants. There is currently ongoing work investigating FTIR in diagnosing malignant pleural mesothelioma and initial results have shown significant spectral differences in this population too. There is very little information regarding the use of FTIR in assessing ascitic fluid. However, despite the technology, it is not available as a bedside point-of-care test for clinicians. The differences and discrimination of the model has not been tested prospectively to determine sensitivity and specificity of the FTIR test. A mobile point-of-care devices that may be able to provide rapid diagnostic results. This study aims to confirm that the spectral changes between malignant and non-malignant samples are present in a UK population in both pleural effusions and ascites.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* A confirmed, clinician made diagnosis of the following (supported by standard accepted diagnostic criteria):
* Malignant pleural effusion: confirmed cancer
* lung cancer
* mesothelioma
* or metastatic cancer
* Non-malignant pleural effusion: effusion confirmed to be caused by alternative diagnosis
* Malignant ascites: confirmed cancer
* Non-malignant ascites: ascites confirmed to be caused by alternative diagnosis
* Willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Unable to comprehend the study
* Unable to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with pleural effusions or ascites will be recruited from outpatient clinics, day units within the hospital and from inpatient wards. Only participants already having a diagnostic or therapeutic procedure as part of their standard medical care will be invited to take part.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
to detect signal difference between malignant and non-malignant pleural effusions | immediately after procedure
  Measured using Fourier transform mid-infrared spectroscopy (FTIR) signal from pleural effusions
To detect a signal difference between malignant and non-malignant ascites | immediately after procedure
  Measured using Fourier transform mid-infrared spectroscopy (FTIR) signal from ascitic fluid
do detect signal difference between malignant and non-malignant pleural effusions | immediately after procedure
  Measured using attenuated Total Reflection Linear Variable Filter (ATR-LVF) spectroscopy signal from pleural effusions
To detect a signal difference between malignant and non-malignant ascites | immediately after procedure
  measured using ttenuated Total Reflection Linear Variable Filter (ATR-LVF) spectroscopy signal from ascitic fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No